CLINICAL TRIAL: NCT02946320
Title: Optimal Predilatation Technique for BVS Implantation
Acronym: OPTI-BVS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cardiology Center Agel (Other)
Responsible Party: Principal Investigator, MUDr. Ivo Varvařovský, Ph.D, Head of Cardiology Center Agel, Cardiology Center Agel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG4201601
Record Dates: First submitted 2016-10-21; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Stenosis
Keywords: PCI, bioabsorbable scaffold
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-compliant balloon (Active Comparator): 15 patients, before BVS implantation is coronary artery stenosis dilated with this type of balloon
  Interventions: Device: Predilatation with non-compliant balloon
- Scoring balloon (Experimental): 15 patients, before BVS implantation is coronary artery stenosis dilated with this type of balloon
  Interventions: Device: Predilatation with scoring balloon (Scoroflex)
- Cutting balloon (Experimental): 15 patients, before BVS implantation is coronary artery stenosis dilated with this type of balloon
  Interventions: Device: Predilatation with cutting balloon (Flextome)

INTERVENTIONS:
Device: Predilatation with non-compliant balloon — Coronary artery stenosis is dilated before BVS implantation with the use of non-compliant balloon (standard procedure). Size and dilatation pressure is done according to OCT measurement of the coronary artery (distal segment / balloon diameter = 1:1)
  Arms: Non-compliant balloon
Device: Predilatation with scoring balloon (Scoroflex) — Coronary artery stenosis is dilated before BVS implantation with the use of scoring balloon. Size and dilatation pressure is done according to OCT measurement of the coronary artery (distal segment / balloon diameter = 1:1)
  Arms: Scoring balloon
Device: Predilatation with cutting balloon (Flextome) — Coronary artery stenosis is dilated before BVS implantation with the use of cutting balloon. Size and dilatation pressure is done according to OCT measurement of the coronary artery (distal segment / balloon diameter = 1:1)
  Arms: Cutting balloon

SUMMARY:
The purpose of this study is to determine the optimal way of predilatation for BVS implantation.

DETAILED DESCRIPTION:
Randomized, single-center study. Forty-five patients with intended BVS implantation will be randomized in ratio of 1:1:1 to different predilatation strategies(non-compliant balloon/Emerge NC™, Boston Scientific, cutting balloon/Flexitome™, scoring balloon/Scoroflex™,Orbus). Predilatation is intended to be done in a vessel:balloon ratio of 1:1. If the device is not able enter the lesion, it will be replaced with a conventional semicompliant balloon with the same predilatation strategy (a vessel:balloon ratio of 1:1) After a successful predilatation, the BVS (Absorb™, Abbott) will be implanted and this procedure will be accomplished by a high pressure postdilatation with a non-compliant balloon (Emerge NC™, BSCI). The MLA of the Absorb stent will be evaluated with optical coherence tomography (OPTIS, St.Jude).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing percutaneous coronary intervention (PCI)
* lesion no more than 25 mm in length with a reference-vessel diameter of 2.5 to 3.75 mm on visual assessment

Exclusion Criteria:

* patients with acurate myocardial infarction (STEMI)
* patients with specific complex lesion features (left main, aorto ostial, bifurcation with side branch ≥ 2 mm in diameter, extreme angulation proximal or within the target lesion, moderate or heavy calcification proximal or within the target lesion, chronic total occlusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Minimal lumen area (MLA) in the BVS (mm2) | Immediately after BVS implantation
  After BVS implantation, optical coherence tomography is used to measure MLA in the scaffold area.

SECONDARY OUTCOMES:
Clinically - driven target vessel revascularization | 12 months after the procedure
  Patient is followed after BVS implantation in 1,6 and 12 months in the outpatient department.
Eccentricity index | Immediately after BVS implantation
  After BVS implantation, optical coherence tomography is used to measure MLA in the scaffold area. Eccentricity index is calculated as minimal luminal diameter divided by maximal luminal diameter in the MLA segment.
Expansion index | Immediately after BVS implantation
  After BVS implantation, optical coherence tomography is used to measure MLA in the scaffold area. Expansion index is calculated as minimal luminal diameter divided by maximal expected diameter of the non-compliant balloon used for high pressure postdilatation.

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Varvařovský, MUDr, Ph.D, Principal Investigator — Cardiology Center AGEL a.s.

IPD SHARING:
Plan to Share IPD: Yes